CLINICAL TRIAL: NCT05252507
Title: Art for Hearts/Black Women's Hearts Paint Night
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Association of Black Cardiologists (ABC) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HM20021891
Record Dates: First submitted 2022-02-14; First posted 2022-02-23 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Stress; Blood Pressure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Paint Night (Experimental)
  Interventions: Behavioral: Paint Night

INTERVENTIONS:
Behavioral: Paint Night — There will be 8 Sessions (4 paint nights and 4 educational sessions alternating weeks). For the painting sessions, participants will paint for 45 minutes and then participate in a combined presentation/discussion session (45 minutes). For the educational sessions, they will attend a 30-minute presentation presented by a researcher on heart health and then have the opportunity to discuss with the researcher and other members of the group (60 minutes).

SUMMARY:
The purpose of this research study is to learn about different techniques that can be used to increase self-reflection, reduce stress, manage high blood pressure in Black women.

DETAILED DESCRIPTION:
The researchers want to know how Black women process stress and cope with it during the pandemic, and if managing stress related through a tailored stress reduction activity/art program affect psychological and blood pressure outcomes over the course of 2 months. It is possible that this information may help people reduce their stress and get treatment for high blood pressure sooner, which can help prevent other heart problems over time.

ELIGIBILITY:
Inclusion Criteria:

* self-identify as African American or black
* have a measured blood pressure (BP) of <140/90 mmHg

Exclusion Criteria:

* Are experiencing cognitive impairment
* Report an untreated psychotic disorder, bipolar disorder, any organic brain syndromes, or substance abuse disorder that the study team believes may result in being a threat to themselves or others
* Report hospitalization for any psychiatric disorder within the past 12 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 20 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2022-10-04 (Actual); Study Completion 2022-10-04 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure | Baseline to 8 weeks
  Participants will take their BP at least once a week (with at least 7 days separating the first and last reading each month) for eight consecutive weeks.
Change in psychological state | Baseline to 8 weeks
  Participants will complete a survey regarding their psychological state at baseline at the conclusion of their 8-week series.

CONTACTS AND LOCATIONS:
Overall Officials: Anika L Hines, PhD, MPH, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No